CLINICAL TRIAL: NCT00533234
Title: ExploR® Modular Radial Head Data Collection
Status: Terminated | Type: Observational
Why Stopped: There was a lack of business need to continue this data collection.
Sponsor: Biomet Orthopedics, LLC (Industry)
Responsible Party: Sponsor
Organization: Zimmer Biomet (Industry)
Other Study IDs: 116-U-001
Record Dates: First submitted 2007-09-20; First posted 2007-09-21 (Estimated); Last update posted 2017-06-21 (Actual); Status verified 2017-06

CONDITIONS: Degenerative Conditions of the Radial Head/Neck; Post-traumatic Conditions of the Radial Head/Neck
Keywords: Elbow fracture; Elbow dislocation; Radial head fracture; Radial neck fracture
MeSH Terms: conditions — Elbow Fractures; Radial Head and Neck Fractures

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: ExploR® Modular Radial Head — The ExploR® Modular Radial Head is a modular head and stem radial head/neck replacement.

SUMMARY:
The purpose of this prospective clinical data collection is to document the performance and clinical outcomes of the ExploR® Modular Radial Head. This data collection effort will document the clinical outcomes of the radial head.

DETAILED DESCRIPTION:
Data collection intervals are:

Pre-operative, Operative, 3 Months Post-op, 1 Year Post-op, 3 Years Post-op, and 5 Years Post-op.

Data collected includes:

Historical data, Operative record, Mayo Clinic Performance Index for the Elbow, Quick DASH Outcome Measure, Complications, Lost to Follow-up, Protocol Deviations, and Radiographic evaluation of elbow and wrist.

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria will be the same as the indications stated in the FDA cleared (510(k) K040611) and (510(k) K051385) labeling for the device.

1. Replacement of the radial head for degenerative or post-traumatic disabilities presenting pain, crepitation, and decreased motion at the radio-humeral and/or proximal radio-ulnar joint with:

   1. Joint destruction and/or subluxation visible on x-ray
   2. Resistance to conservative treatment
2. Primary replacement after fracture of the radial head
3. Symptomatic sequelae after radial head resection
4. Revision following failed radial head arthroplasty

The device is intended for single use with or without bone cement.

Modular Radial Head replacement prostheses have received FDA clearance for cemented and non-cemented application.

Patient selection factors to be considered include: 1) need to obtain pain relief and improve function, 2) ability and willingness of the patient to follow instructions, including control of weight and activity levels, 3) a good nutritional state of the patient, and 4) the patient must have reached full skeletal maturity.

Exclusion Criteria:

The exclusion criteria will be the same as the contraindications stated in the FDA cleared labeling (510(k) K040611) and (510(k) K051385) for the device. These contraindications include:

Absolute contraindications:

1. Infection
2. Sepsis
3. Osteomyelitis

Relative contraindications:

1. Uncooperative patient or patient with neurologic disorders who is incapable or unwilling to follow directions
2. Osteoporosis
3. Metabolic disorders which may impair bone function
4. Osteomalacia
5. Distant foci of infections which may spread to the implant site
6. Rapid joint destruction, marked bone loss or bone resorption apparent on roentgenogram.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will be implanted with the ExploR® Modular Radial Head.
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2009-12; Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Mayo Clinic Performance Index for The Elbow, Quick DASH Outcome Measure, Radiographic Evaluation | 5 years

SECONDARY OUTCOMES:
Revisions, Complications, Adverse Events | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Ken Beres, MD, Principal Investigator — Biomet Orthopedics, LLC
Locations (1):
- Biomet Orthopedics, LLC, Warsaw, Indiana, United States